CLINICAL TRIAL: NCT05908279
Title: Flexible Control of Gait in Parkinson Disease: Effect of Task Instruction on the Exploitation of Redundancy in Speed Control.
Brief Title: Gait Control in Parkinson Disease
Acronym: GAIT-PD
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: GAIT-PD
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD: Patients with Parkinson's disease
  Interventions: Other: Walking test; Other: Disease assessement
- Control: Healthy volunteers
  Interventions: Other: Walking test

INTERVENTIONS:
Other: Walking test — Walk with and without a metronome
Other: Disease assessement — Disease stage assessed by a doctor
  Groups: PD

SUMMARY:
Previous work has shown that a statistical property of gait characterised by long-range autocorrelation functions is altered in Parkinson disease (PD). On the other hand it has been suggested that the same property is linked to the ability in healthy humans to co-regulate the amplitude and cadence of strides towards maintaining a constant speed. Here the investigators want to better understand why it is altered in PD by measuring the transitions between gait instructed by a metronome, and gait without metronome. The experimental conditions will allow the comparisons between these transitions across PD and healthy groups of volunteers, and assess differences based on statistical and computational modelling. The link with potential freezing episodes will also be studied to assess whether the statistical determinants of gait control in this population can be used as a proxy or predictor of the occurence of freezing episodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients and volunteers able to walk for 20mins and without other neurological disorders.

Exclusion Criteria:

* Patients or volunteers unable to walk for 20mins and with other neurological disorders.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One group of volunteers with previous diagnosis of Parkinson disease and one group of age and sex matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Stride cadence | Measured during the entire experiment (an average of 4.5 years)
  Time between two consecutive heel strikes. Units are seconds.
Stride amplitude | Measured during the entire experiment (an average of 4.5 years)
  Distance between two consecutive heel strikes. Units are meters.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Crevecoeur, Study Director — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No